CLINICAL TRIAL: NCT02339129
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Determine the Dosing Interval, Efficacy, and Safety of SST-0225, a Topical Ibuprofen Cream, in the Treatment of Delayed Onset Muscle Soreness (DOMS)
Brief Title: Dosing Interval Study of SST-0225 Topical Ibuprofen Cream in the Treatment of Delayed Onset Muscle Soreness
Acronym: DIS DOMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Strategic Science & Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SST0225-US-111-001A
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Delayed Onset Muscle Soreness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SST-0225 (Experimental): Subjects will be treated with IP for 48 hours. While on-site, subjects will apply the first dose of IP at 0 hours, the second dose upon request (PRN), and all subsequent doses every 5 (±1) hours, up to a maximum of 6 doses in 24 hours. After subjects complete their 24 hour post first dose VAS pain/soreness on movement assessment, they will be released from the clinic and will continue outpatient treatment for the remaining 24 hours. While off-site subjects will dose every 5 (±1) hours, not to exceed 6 doses in 24 hours.
  Interventions: Drug: SST-0225
- Placebo (Placebo Comparator): Subjects will be treated with IP for 48 hours. While on-site, subjects will apply the first dose of IP at 0 hours, the second dose upon request (PRN), and all subsequent doses every 5 (±1) hours, up to a maximum of 6 doses in 24 hours. After subjects complete their 24 hour post first dose VAS pain/soreness on movement assessment, they will be released from the clinic and will continue outpatient treatment for the remaining 24 hours. While off-site subjects will dose every 5 (±1) hours, not to exceed 6 doses in 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SST-0225 — SST-0225 is a cream formulation for topical application. Each 5.4 g dose is formulated to topically deliver 400 mg of ibuprofen. The cream contains sodium ibuprofen and various salts.
  Other Names: Topical Ibuprofen Cream
  Arms: SST-0225
Drug: Placebo — Placebo IP will be the same vehicle as SST-0225 vehicle without the active ingredient, ibuprofen. It will be matched in appearance, smell, consistency, and color to SST-0225 topical ibuprofen cream.
  Arms: Placebo

SUMMARY:
This is a Phase 2, prospective, randomized, dual-center, double-blind, placebo-controlled, parallel-group study designed to determine the dosing interval, efficacy and safety of SST-0225 (5.4 grams, applied up to 6 times in 24 hours, over a 48-hour dosing period) for the treatment of pain associated with DOMS.

DETAILED DESCRIPTION:
This is a Phase 2, prospective, randomized, dual-center, double-blind, placebo-controlled, parallel-group study designed to determine the dosing interval, efficacy and safety of SST-0225 (5.4 grams, applied up to 6 times in 24 hours, over a 48-hour dosing period) for the treatment of pain associated with DOMS.

As part of the screening process, in the evening of Day -2, eligible subjects will undergo an exercise regimen designed to induce DOMS in the elbow flexor of the non-dominant arm (see Section 11). 36 (±2) hours following the exercise regimen, subjects will return to the clinic and be evaluated for eligibility into the active treatment phase of the study. Eligible subjects who experience a sufficient level of pain 36 (± 2) hours after exercise will be randomized to receive either SST-0225 or placebo.

For the first 24 hour dosing period, the subject will remain in the clinic (on-site). Subjects will apply the first dose of Investigational Product (IP) at randomization (0 hours) and a second dose upon request (PRN or as needed). All subsequent doses will be applied every 5 (±1) hours. The total number of doses shall not exceed 6 in this first 24 hour period. Subjects will also not be allowed to take any rescue medication during the first 24 hour dosing period.

Subjects will complete the Visual Analog Scale (VAS) pain/soreness on movement assessments at the following time points while on-site the first 24 hours: 0 (prior to first dose of IP), 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16, and 24 hours post first dose of IP and immediately prior to the second dose of IP. All assessments must be completed unless the subject is asleep. Subjects will be restricted to a maximum of 8 hours of sleep in order to limit the number of missing VAS pain/soreness on movement assessments due to sleep. Immediately upon wakening on Day 2, subjects will be instructed to apply a dose of IP unless it has been less than 5 (±1) hours since their last dose of IP.

After subjects complete their 24 hour VAS pain/soreness on movement assessment, they will be released from the clinic and will continue outpatient treatment for the second 24 hour dosing period.

During the second 24 hour dosing period (24-48 hours post first dose of IP), the subject will be away from the clinic (off-site) and will apply the IP every 5 (±1) hours. The total number of doses shall not exceed 6 doses in this second 24 hour period. Rescue medication will be made available to subjects during this second 24 hour period. During this second 24 hour period, subjects will complete the VAS pain/soreness on movement assessment prior to each IP dose and at 1 hour post each dose of IP.

Refer to the Schedule of Evaluations in Appendix A (on-site evaluations) and Appendix B (off-site evaluations) for details regarding the timing of study procedures.

ELIGIBILITY:
Healthy male and female subjects between 16 and 65 years of age.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
SPID24 (calculated by summing the time weighted VAS pain/soreness on movement assessment differences from baseline) | First 24 hours after first dose
  The primary efficacy endpoint will be the time weighted summed pain/soreness intensity difference from baseline VAS pain/soreness on movement assessments over the first 24 hours (SPID24) following the first application of IP on Day 1. SPID24 will be calculated by summing the time weighted VAS pain/soreness on movement assessment differences from baseline (pre-dose on Day 1) to 24 hours (using actual reported VAS assessment times) post first dose of IP on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Howard I Schwartz, MD, Principal Investigator
Locations (2):
- United States (2):
  - Site #201, South Miami, Florida
  - Site #202, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: Undecided